CLINICAL TRIAL: NCT00465322
Title: Effect of Fluvastatin on Top of Clopidogrel and Aspirin in Patients After DES Implantation on Platelet Aggregation
Acronym: EFA-1
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Other Study IDs: 1101
Record Dates: First submitted 2007-04-23; First posted 2007-04-25 (Estimated); Last update posted 2007-04-25 (Estimated); Status verified 2007-04

CONDITIONS: Drug-Interactions
MeSH Terms: interventions — Fluvastatin

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: fluvastatin

SUMMARY:
The purpose of the study was to determine the influence of fluvastatin and atorvastatin on platelet aggregation in patients treated with aspirin and plavix after coronary stenting. We hypothezied a positive effect of fluvastatin on platelet aggregation levels.

DETAILED DESCRIPTION:
1. Introduction Coronary stent implantation is performed in more than 80 % of all coronary interventions. The use of stents has significantly reduced re-stenosis rate in revascularization in comparison with conventional balloon angioplasty. To prevent stent thrombosis dual antiplatelet therapy with acetylsalicylic acid and clopidogrel (ADP-receptor antagonist) is routinely used (1).

   Previous studies reported a drug interaction between clopidogrel and several statins (e.g. atorvastatin, simvastatin) and described a dose-dependent inhibition of the effect of clopidogrel on platelet aggregation. This drug interaction is thought to be due to the fact that both drugs (clopidogrel and atorvastatin/simvastatin) are metabolized by cytochrome P450 3A4 (2, 3). In contrast to atorvastatin and simvastatin, fluvastatin is mainly metabolized by cytochrome P450 2C9. Metabolization of clopidogrel is mandatory for effective platelet inhibition. Since all patients after coronary stent implantation are treated with clopidogrel and over 80 % of patients with coronary heart disease receive a statin the question whether there is a drug-drug interaction is of great importance.

   In a previous trial we observed a beneficial effect of fluvastatin on platelet inhibition on top of aspirin and Clopidogrel (4). There was a further reduction of platelet aggregation of approximately 10%, whereas atorvastatin or pravastatin had no effect or even slightly increased platelet aggregation.
2. Aim

   The purpose of the present study is 1) to determine a beneficial effect of fluvastatin on platelet aggregation in comparison with atorvastatin in patients with stable coronary artery 2) to assess a potential drug-drug interaction of Clopidogrel and atorvastatin .
3. Patients and Methods Approximately 100 patients are included in the present study. All patients undergo coronary stent implantation with a drug eluting stent. The first measurement of platelet aggregation under aspirin and clopidogrel treatment (loading dose 600mg) is set to be between 12 and 24 hours after the administration of the loading dose of clopidogrel. Any statin treatment will be stopped for 2 weeks (washout phase for statin treatment before study inclusion) after the PCI. After 2 weeks second platelet aggregation under the treatment with ASA and clopidogrel and randomization to fluvastatin 80mg and atorvastatin 40mg per day in addition to the dual antiplatelet therapy. Third measurement 1 month later and crossover of statin treatment for another month. End of the study with a forth measurement of platelet aggregation.

Clinical follow-up (MACE) 2.5, 6 and 12 months after inclusion.

Measured variables:

1. Platelet aggregation will be assessed by the following method:

   · APACT-4 aggregometer (Endothell, Switzerland, induced by 5, 20 µmol ADP and 0.5mg/ml arachidonic acid) (5).
2. Blood analysis: Blood smear, coagulation parameters, lipid profile, liver enzyme, creatinkinase, homocysteine, hs-CRP, BNP

Sample size justification: It is estimated that 50 patients per treatment group will provide 99% power to achieve a 10% difference in platelet aggregation (± 10 standard deviation).

4. Study Design and Duration

Duration: 12 months, 2.5 months for assessment of platelet aggregation Primary endpoint: platelet aggregation after 2.5 months Secondary endpoint: MACE after 12 month

5. Inclusion Criteria

* all patients with stent implantation followed by treatment with aspirin and clopidogrel
* routinely treated with acetylsalicylic 100 mg/day

  6. Exclusion Criteria
* acute coronary syndrome
* use of a GPIIb/IIIa inhibitor
* allergy to acetylsalicylic acid, clopidogrel, statins
* elevated liver enzymes (> 3 x norm value)
* muscle myopathy
* active liver disease
* recent gastrointestinal bleeding (< 3 months)
* known platelet dysfunction or abnormal platelet count
* pregnancy
* indication for treatment with non-steroidal drugs
* indication for long-term treatment with a drug metabolized by cytochrome p450 3A4 or 2C9

  7. Literature
  1. Berger, P.B., et al., Clopidogrel versus ticlopidine after intracoronary stent placement. J Am Coll Cardiol, 1999. 34(7): p. 1891-4.
  2. Lau, W. C., L. A. Waskell, et al. (2003). "Atorvastatin reduces the ability of clopidogrel to inhibit platelet aggregation: a new drug-drug interaction." Circulation 107(1): 32-7.
  3. Clarke TA, Waskell LA. The metabolism of clopidogrel is catalyzed by human cytochrome P450 3A and is inhibited by atorvastatin. Drug Metab Dispos 2003;31(1):53-9
  4. Wenaweser P., et al. Do Statins Interfere With the Antiaggregatory Effect of Clopidogrel in Patients With Stent Thrombosis ? Abstract presentation Swiss Cardiac Society, June 2005, Lausanne
  5. McKenzie ME, Gurbel PA, Levine DJ, Serebruany VL. Clinical utility of available methods for determining platelet function. Cardiology. 1999;92(4):240-7. Review

ELIGIBILITY:
Inclusion Criteria:

* all patients with stent implantation followed by treatment with aspirin and clopidogrel
* routinely treated with acetylsalicylic 100 mg/day

Exclusion Criteria:

* acute coronary syndrome
* use of a GPIIb/IIIa inhibitor
* allergy to acetylsalicylic acid, clopidogrel, statins
* elevated liver enzymes (> 3 x norm value)
* muscle myopathy
* active liver disease
* recent gastrointestinal bleeding (< 3 months)
* known platelet dysfunction or abnormal platelet count
* pregnancy
* indication for treatment with non-steroidal drugs
* indication for long-term treatment with a drug metabolized by cytochrome p450 3A4 or 2C9

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100

CONTACTS AND LOCATIONS:
Overall Officials: Otto M Hess, Prof., Principal Investigator — Cardiology University Hospital Bern; Peter Wenaweser, MD, Principal Investigator — Cardiology University Hospital Bern
Locations (1):
- Cardiology University Hospital, Bern, Switzerland

REFERENCES:
- [Derived] Wenaweser P, Eshtehardi P, Abrecht L, Zwahlen M, Schmidlin K, Windecker S, Meier B, Haeberli A, Hess OM. A randomised determination of the Effect of Fluvastatin and Atorvastatin on top of dual antiplatelet treatment on platelet aggregation after implantation of coronary drug-eluting stents. The EFA-Trial. Thromb Haemost. 2010 Sep;104(3):554-62. doi: 10.1160/TH09-11-0765. Epub 2010 Jul 20. PMID 20664903